CLINICAL TRIAL: NCT05114473
Title: Educational Program Interventions for Patients Suffering From Persistent Pelvic Pain and Their Effects Over Pain and Functionality. A Multi-centered Randomized Clinical Trial.
Brief Title: Efficacy of Pain Neuroscience Education in Genito-Pelvic Pain/Penetration Disorder. A Randomized Controlled Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Borja Pérez-Domínguez, Associate Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UV-INV_ETICA-1741806
Record Dates: First submitted 2021-10-25; First posted 2021-11-10 (Actual); Results first posted 2024-05-23 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Pain; Dysfunction Sexual
MeSH Terms: conditions — Pain; Sexual Dysfunction, Physiological

STUDY DESIGN:
Intervention Model Description: Two groups receiving intervention and one serving as control
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Due to the nature of the intervention, participants can't be blinded to allocation, but are strongly inculcated not to disclose the allocation their status at the follow up assessments. Care providers will be different from outcome assessors and will be both blinded by an external investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Workshops (Experimental): This group will attend face-to-face workshops were the educational program will be developed. These workshops will be available in several sites, and specific care providers will be assigned for each of these sites.
  Interventions: Other: Workshops
- Online-accessed material (Experimental): This group will be granted online access to a platform were the educational program will be uploaded. They will be given autonomy regarding when to enter the platform and view the content.
  Interventions: Other: Online-accessed material
- Control group (No Intervention): This group will initially no recieve an intervention and will serve as a control group.

INTERVENTIONS:
Other: Workshops — Several face-to-face workshops given by a researcher
  Arms: Workshops
Other: Online-accessed material — Access to a website containing the educational program
  Arms: Online-accessed material

SUMMARY:
Patients suffering pelvic persistent pain deal with significant pain that affects their quality of life. Often, conservative treatment interventions are scarce for these patients and are therefore not considered. Education has been developed as a relevant tool in the treatment of patients who suffer from chronic pain or any other pain processing alterations, and has the potential to become a powerfull treatment alternative.

DETAILED DESCRIPTION:
In this intervention, the effects of implementing educational programs in patients suffering from pelvic persistent pain will be assessed.

Patients with pelvic persistent pain have both problems directly related with their pain and other issues that appear derived from suffering pain over a determined period, such as alterations in the sexuality or overall quality of life. Facing these patients is a challenge for professionals, and many can't find the treatment that properly fits the patient's clinical presentation.

Education, and educating patients on their problem, is an exponentially growing alternative used in Physical Therapy involving patients who suffer from a dysfunctional pain, chronic pain, or any kind of pain presentation that affects the patient's well-being.

This study will assess firstly if the implementation of a pain-related education program is relevant in the treatment of pelvic persistent pain, and will further observe which modality (presential workshops or online-accessed material) is the most effective involving adherence and improvement.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years-old suffering from dyspareunia for more than 3 months

Exclusion Criteria:

* Patients suffering from a previous medical condition that explains logically the presence of pain

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Valencia, Spain

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Workshops | Online-accessed Material | Control Group
Started | 18 | 29 | 22
Completed | 16 | 27 | 22
Not Completed | 2 | 2 | 0
Not completed — Lost to Follow-up | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Workshops | Online-accessed Material | Control Group | Total
Number analyzed (Participants) | 18 | 29 | 22 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (13.2) | 31.6 (6.9) | 33.0 (9.1) | 32.8 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 29 | 22 | 69
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale
Description: Pain intensity assessment instrument. Minimum value 0, maximum value 10. Higher scores mean worse outcome
Time Frame: Baseline to week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Workshops | Online-accessed Material | Control Group
Number analyzed (Participants) | 16 | 27 | 22
score on a scale
  Pre | 5.3 (2.5) | 5.8 (2.0) | 5.1 (1.8)
  Post | 3.8 (2.4) | 4.9 (2.5) | 4.9 (2.2)

2. Secondary Outcome: Pain Catastrophizing Scale
Description: Instrument developed quantify an individual's pain experience. Minimum value 0, maximum value 52. Higher scores mean worse outcome
Time Frame: Baseline to week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Workshops | Online-accessed Material | Control Group
Number analyzed (Participants) | 16 | 27 | 22
score on a scale
  Pre | 25.2 (12.7) | 28.0 (10.4) | 22.4 (7.5)
  Post | 18.9 (12.6) | 20.4 (11.5) | 25.3 (8.2)

3. Secondary Outcome: Survey of Pain Attitudes
Description: Instrument to understand the pain-related beliefs of your chronic pain patients. Minimum value 0, maximum value 285. Higher scores mean better results
Time Frame: Baseline to week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Workshops | Online-accessed Material | Control Group
Number analyzed (Participants) | 16 | 27 | 22
score on a scale
  Pre | 45.1 (10.6) | 49.6 (13.1) | 52.4 (13.0)
  Post | 45.2 (14.5) | 50.9 (14.8) | 52.4 (13.6)

4. Secondary Outcome: Female Sexual Function Index
Description: Inventory designed to assess female sexual function. Minimum value 2, maximum value 36. Higher scores mean better functioning
Time Frame: Baseline to week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Workshops | Online-accessed Material | Control Group
Number analyzed (Participants) | 16 | 27 | 22
score on a scale
  Pre | 18.9 (7.8) | 19.1 (7.3) | 19.5 (7.1)
  Post | 21.0 (9.5) | 20.8 (8.1) | 18.4 (9.3)

ADVERSE EVENTS:
Time Frame: Adverse event data was not collected.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Workshops | Online-accessed Material | Control Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
No limitations or caveats were found

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT05114473/Prot_SAP_000.pdf